CLINICAL TRIAL: NCT01070797
Title: Administration of Rapidly Generated Multivirus-specific Cytotoxic T-Lymphocytes for the Prophylaxis and Treatment of EBV, CMV, and Adenovirus Infection Post Allogeneic Stem Cell Transplant (VIRAGE)
Brief Title: Administration of Rapidly Generated Multivirus-specific Cytotoxic T-Lymphocytes (VIRAGE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor of Pediatrics-Hem-Onc Cell & Gene, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26374-VIRAGE; VIRAGE (Other: Baylor College of Medicine)
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Adenovirus Infection; Epstein-Barr Virus Infections; Cytomegalovirus Infections; Stem Cell Transplant
Keywords: Epstein-Barr virus; CTL; cytotoxic T Lymphocytes; CMV; Adenovirus Infection; viral infection; hematopoietic stem cell transplantation
MeSH Terms: conditions — Adenoviridae Infections; Epstein-Barr Virus Infections; Cytomegalovirus Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A is for CMV seropositive donors.
  Interventions: Biological: Multi-virus Specific T cells
- Group B (Experimental): Group B is for CMV seronegative donors.
  Interventions: Biological: Multi-virus Specific T cells

INTERVENTIONS:
Biological: Multi-virus Specific T cells — Subjects will receive Multivirus specific T cells on one of the following dose levels:
  Level One: 5 x 10^6 rCTLs/m2
  Level Two: 1 x 10^7 rCTLs/m2
  Level Three: 2 x 10^7 rCTLs/m2
  Level Four: 5 x 10^7 rCTLs/m2
  If a patient has a partial response (as defined by a 50% fall in viral load) or receives medication (such as steroids) which may affect the persistence or function of the infused CTL they are eligible to receive up to 2 additional doses at the same initial dose. The minimum time between additional doses is 28 days.

SUMMARY:
Patient's on this protocol have a type of blood cell cancer, other blood disease or a genetic disease and have received a stem cell transplant. The donor of the stem cells was either a brother or sister, another relative, or a closely matched unrelated donor. The patient is being asked to participate in this study which tests if blood cells from the donor that have been grown in a special way, can prevent or be an effective treatment for early infection by three viruses - Epstein Barr virus (EBV), cytomegalovirus (CMV) and adenovirus.

Adenovirus is a virus that usually causes symptoms of a common cold, but can cause serious life-threatening infections in patients who have weak immune systems. It can affect the lungs and cause very serious pneumonia, and can also damage the gut, liver, pancreas and eyes.CMV can also cause serious infections in patients with weak or suppressed immune systems. It usually affects the lungs, causing a very serious pneumonia, but it can also affect the gut, the liver and the eyes. Approximately 2/3 of normal people harbor this virus in their body. In healthy people CMV rarely causes any problems because the immune system can keep it under control, but after a transplant, the risk of developing CMV disease is much higher because the immune system is so weak. EBV is the virus that causes glandular fever. It is also a life long infection like CMV that is normally controlled by the immune system. When immunity is weak, the virus can become active and cause fevers, enlarged lymph nodes and sometimes a type of cancer called lymphoma.

Investigators want to see if a kind of white blood cell called T lymphocytes (T cells)can be used to prevent and treat adenovirus, CMV and EBV in the early stages of reactivation or infection. T cells have been grown from the patient's stem cell donor in the laboratory in a way that will train them to recognize the virus and control it when they are given after a transplant. This treatment with specially trained T cells (also called CTLs) has had activity against these viruses in previous studies and in this study investigators want to see if they still have activity when they are made in a simpler and faster way. These donor-derived multivirus-specific special cell lines are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to evaluate whether donor-derived multivirus-specific special cell lines are safe and can control three viruses: EBV, CMV and adenovirus.

DETAILED DESCRIPTION:
Blood has been previously taken from the patient and the donor to make the cells.

To make the special cell line, special blood cells called dendritic cells (DCs)were made first from the donor blood. Then, a specially produced gene called a plasmid that carries the adenovirus, CMV, and EBV genes was introduced into the dendritic cells. Dendritic cells with these new genes are then mixed with T cells to stimulate them. This stimulation trains the donor T cells to kill cells that are infected with CMV, EBV, and adenovirus. Once a sufficient numbers of T cells were made, they were tested to make sure they killed the patient's cells infected with these viruses, but not the patient's normal cells, and were frozen.

If the donor has never been infected with CMV, the CTLs made for the patient may not have activity against a CMV infection. If these donor CTLs show no activity against CMV infection, the cells will not be given.

The patient may receive Benadryl (diphenhydramine) and Tylenol (acetaminophen). Then, the donor's special cells will be thawed and injected into the patient's intravenous line. After the patient receives the cells, the levels of these three viruses in the patient's blood will be monitored. Investigators will also take blood to see how long the T cells given to the patient are lasting in the patient's body.

If the special cell infusion has helped the infection or if the patient has had a treatment (for example with steroid drugs) that might have destroyed the T cells that were given to them, then the patient is allowed to receive up to 2 more doses of the cells.

The patient will continue to be followed by his/her transplant doctors after the injection. The patient will either be seen in the clinic or contacted by a research nurse to follow up for this study every week for 6 weeks then at 8 weeks, and 3, 6, and 12 months. The patient may have other visits for standard care.

The patient will also have regular blood tests done to follow counts and the viral infection. To learn more about the way the T cells are working in the patient's body, up to an extra 30-40 ml (6-8 teaspoons) of blood will be taken before the infusion and then at 1, 2, 4, 6, and 8 weeks and 3 months. Blood should come from the central intravenous line, and should not require extra needle sticks. Total time participation for this study will be 1 year.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients will be eligible following any type of allogeneic transplant to receive CTLs as prophylaxis or for early reactivations as defined below.

1. Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cells.
2. Prophylaxis for patients at risk of CMV, adenovirus or EBV infection (for Phase 2 portion only). In the phase 1 portion patients must meet criteria in 3 below.
3. Early treatment of reactivation or infection which is defined for each virus as below:

   1. CMV: CMV antigenemia is monitored at least weekly post transplant. Early reactivation is defined at CMV antigenemia with less than 10 leucocytes positive. If any patient develops CMV antigenemia (with greater than 10 leukocytes positive) or clinical evidence of CMV infection (defined as the demonstration of CMV by biopsy specimen from visceral sites (by culture or histology) either pre or after CTL infusions, standard treatment with Ganciclovir, and/or Foscarnet and Immunoglobulins will be initiated. Patients may receive CTLs for antigenemia or elevated PCR without visceral infection.
   2. Adenovirus: Adenovirus infection will be defined as the presence of adenoviral positivity as detected by PCR or culture from ONE site such as stool or blood or urine or nasopharynx. Adenovirus disease will be defined as the presence of adenoviral positivity as detected by culture from more than two sites such as stool or blood or urine or nasopharynx. In patients who meet the criteria for disease Cidofovir may be added unless the subject could not tolerate this agent due to nephrotoxicity. Patients may receive CTLs for elevated PCR in blood or stool.
   3. EBV EBV-LPD is defined according to recent guidelines as proven EBV-LPD defined by biopsy or probable EBV-LPD defined as an elevated EBV DNA level associated with clinical symptoms (adenopathy or fever or masses on imaging) but without biopsy confirmation. Patients with EBV DNA reactivation only defined as EBV DNA levels > 1000 copies/ug may also receive CTLs on study. Patients with proven or probable EBV-LPD should also receive Rituxan
4. Early treatment may be given to eligible patients with a single or multiple infections. Patients with multiple infections with one reactivation and one controlled infection are eligible to enroll.
5. Patient with a CMV seronegative donor may only receive CTLs for a CMV reactivation in the dose escalation phase if the line has activity against CMV.
6. Clinical status at enrollment to allow tapering of steroids to less than 0.5 mg/kg/day prednisone.
7. Karnofsky/Lansky score of 50 or greater
8. ANC greater than 500/µL.
9. Bilirubin 2x upper limit normal or less
10. AST 3 x normal or less
11. Serum creatinine 2 x upper limit normal or less
12. HgB >8.0
13. Pulse oximetry of > 90% on room air
14. Available multi-virus-specific cytotoxic T lymphocytes
15. Negative pregnancy test in female patients if applicable (childbearing potential who have received a reduced intensity conditioning regimen).
16. Written informed consent and/or signed assent line from patient, parent or guardian.

DONOR ELIGIBILITY: The donor for the CTL product will be the same donor who donated the allogeneic product for the patient's transplant. These donors for allogeneic (i.e. HLA matched or mismatched related or unrelated) stem cell transplants will have fulfilled eligibility for and consented to stem cell donation as per the stem cell transplant program's standard operating procedures.

EXCLUSION CRITERIA:

Exclusion Criteria for initial CTL and for subsequent infusions:

1. Patients receiving ATG, or Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of screening for enrollment.
2. Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.

   Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
3. Patients who have received donor lymphocyte infusion (DLI) within 28 days.
4. Patients with active acute GVHD grades II-IV.
5. Active and uncontrolled relapse of malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Assessment of dose limiting toxicity in subjects receiving rapidly-generated donor-derived multivirus-specific CTLs | 42 days
  Safety and toxicity outcomes including DLTs, GvHD, clinical signs of viral infections, secondary graft failure and laboratory measurements will be summarized using descriptive statistics for each dose level (frequency table, means, standard deviations, medians and ranges).
Determine the effect of rCTL infusion on viral load | 1 year
  Primary endpoint for the phase II portion of the study is antiviral efficacy, and is whether the institution of additional antiviral therapy post rCTL is needed.

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Gerdemann U, Katari UL, Papadopoulou A, Keirnan JM, Craddock JA, Liu H, Martinez CA, Kennedy-Nasser A, Leung KS, Gottschalk SM, Krance RA, Brenner MK, Rooney CM, Heslop HE, Leen AM. Safety and clinical efficacy of rapidly-generated trivirus-directed T cells as treatment for adenovirus, EBV, and CMV infections after allogeneic hematopoietic stem cell transplant. Mol Ther. 2013 Nov;21(11):2113-21. doi: 10.1038/mt.2013.151. Epub 2013 Jun 20. PMID 23783429